CLINICAL TRIAL: NCT05005975
Title: A Phase 3, Multicenter, Open-label, Long-term, Extension Study to Evaluate Safety and Tolerability of Oral Dersimelagon (MT-7117) in Subjects With Erythropoietic Protoporphyria (EPP) or X-Linked Protoporphyria (XLP)
Brief Title: Extension Study to Evaluate Safety and Tolerability of Oral Dersimelagon (MT-7117) in Subjects With Erythropoietic Protoporphyria (EPP) or X-Linked Protoporphyria (XLP)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-7117-A-301; jRCT2041210146 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2021-001831-17 (EudraCT Number)
Record Dates: First submitted 2021-07-28; First posted 2021-08-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: EPP; XLP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dersimelagon 200mg (Experimental)
  Interventions: Drug: MT-7117

INTERVENTIONS:
Drug: MT-7117 — MT-7117
  Other Names: Dersimelagon

SUMMARY:
To evaluate the long-term safety and tolerability of oral dersimelagon.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* 1. Subjects provided written informed consent to participate. For adolescent subjects, both adolescent assent and parental consent will be provided.
* 2. Subjects who have completed: MT-7117-G01 (completed through Week 58 [Visit 12]) or, MT-7117-A-302 (completed through Week 58 [Visit 10]) or, MT-7117-A-301 (completed EOT - Week 104 or Week 130) according to protocol amendment 1 or 2.
* 3. Subjects are willing and able to travel to the study sites for all scheduled visits.
* 4. In the Investigator's opinion, subject can understand the nature of the study and any risks involved in participation, and is willing to cooperate and comply with the protocol restrictions and requirements (including travel).
* 5. Female subjects who are non-lactating and have a negative urine pregnancy test at baseline visit prior to receiving the first dose of study drug.
* 6. Female subjects of childbearing potential and male subjects with partner of childbearing potential must agree to use 2 effective methods of contraception including barrier method (especially for female subjects, one method must be highly effective method)

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

A subject will NOT be eligible for this study if ANY of the following criteria apply:

* 1. History or presence of photodermatoses other than EPP or XLP.
* 2. Presence of clinically significant hepatobiliary disease at Screening, determined as clinically significant by the Investigator.
* 3. Subjects with AST, ALT, ALP ≥ 3.0 × upper limit of normal (ULN) or TB > 1.5 × ULN at Screening. The TB level of > 1.5 × ULN listed in this exclusion criteria may not be applicable to subjects with a documented medical history of Gilbert's syndrome. Please consult with the Sponsor for eligibility of subjects with elevated levels due to Gilbert's syndrome.
* 4. Subjects with or having a history (in the last 2 years) of excessive alcohol intake in the opinion of the Investigator.
* 5. History of melanoma.
* 6. Presence of squamous cell carcinoma, basal cell carcinoma, or other malignant skin lesions. Any suspicious lesions or nevi will be evaluated. If the suspicious lesion or nevi cannot be resolved through biopsy or excision, the subject will be excluded from the study.
* 7. History or presence of psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation and/or safety of the subjects.
* 8. Presence of clinically significant acute or chronic renal disease based upon the subject's medical records including hemodialysis; an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 as calculated by the CKD-EPI creatinine equation (2009) for adults and by the Schwartz creatinine equation for adolescents (2009). MDRD can be used for adults per local recommendations.
* 9. Presence of any clinically significant disease or laboratory abnormality which, in the opinion of the Investigator, can interfere with the study objectives and/or safety of the subjects.
* 10. Female subjects who are pregnant, lactating, or intending to become pregnant during the study.
* 11. Treatment with phototherapy or afamelanotide within 3 months before baseline (Visit 2 or Re-entry Visit 2).
* 12. Treatment with cimetidine or antioxidant agents at doses which, in the opinion of the Investigator, may affect study endpoints (including but not limited to beta-carotene, cysteine, pyridoxine) within 4 weeks before baseline (Visit 2 or Re-entry Visit 2).
* 13. Chronic treatment with opioids, ketamine, or medical formulations or derivatives of cannabis within 4 weeks before baseline (Visit 2). Note: This exclusion criterion may not be applicable to subjects at Re-entry Visits. Acute use of scheduled analgesics more than 3 months before baseline (Visit 2) is allowed.
* 14. Treatment with any drugs or supplements which, in the opinion of the Investigator, can interfere with the objectives of the study or safety of the subjects.
* 15. Previous treatment with any investigational agent other than dersimelagon within 12 weeks before Screening OR 5 half-lives of the investigational product (whichever is longer).
* 16. History of any hypersensitivity to the active ingredient and/or excipients (lactose monohydrate, hydroxypropyl cellulose, carmellose calcium, magnesium stearate, hypromellose, titanium dioxide, talc, polyethylene glycol, iron oxide yellow, iron oxide red, and iron oxide black).
* 17. Subjects who are unable to swallow tablets or have diseases significantly affecting the gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* 18. Using the following drugs (including but not limited to) within 1 week of baseline (Visit 2 or Re-entry Visit 2):

  1. Drugs known to be predominantly metabolized by cytochrome P450 (CYP) 3A4 with a narrow therapeutic index for which elevated plasma concentrations are associated with clinical safety concern or significant medical events.
  2. Drugs that are known substrates of P-glycoprotein (P-gp), breast cancer resistance protein (BCRP), organic anion transporting polypeptide (OATP)1B1, or OATP1B3 for which elevated plasma concentrations are associated with significant medical events.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Treatment emergent adverse events (TEAEs) (including serious adverse events [SAEs] and adverse events of special interest [AESIs]). | up to 66 further months
  Vital signs (blood pressure, respiratory rate, pulse rate, and body temperature), Clinical laboratory examinations (hematology, coagulation, biochemistry, urinalysis, and others), 12-lead electrocardiogram (ECG) parameters (Mean Heart Rate, PR Interval, QRS Duration, QT interval, QTcB and QTcF) will be assessed.
Number of patients with abnormal Physical examination data | up to 66 further months
  Physical examination consists of assessment of abdominal, respiratory, cardiovascular, general appearance, and others.
Number of patients with Nevi appearance | up to 66 further months

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (51):
- United States (15):
  - Marvel Clinical Research, LLC, Huntington Beach, California
  - University of California at San Francisco - CSF Porphyria Center, San Francisco, California
  - University Of Miami School Of Medicine, Center For Liver Diseases, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - MetroBoston Clinical Partners, LLC, Brighton, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Kansas City Research Institute, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai (ISSMS)-The Mount Sinai Hospital (MSH), New York, New York
  - Wake Forest University Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Medical Branch (UTMB), Galveston, Texas
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Wesley Medical Research, Brisbane, Queensland
  - Royal Melbourne Hospital (RMH), Parkville, Victoria
- University Multi-Profile Hospital for Active Treatment (UMHAT) St. Ivan Rilski, Sophia, Belgium
- University of Alberta Hospital, Edmonton, Alberta, Canada
- Institute for Clinical and Experimental Medicine - IKEM, Prague, Czechia
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint - Andre, Bordeaux
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Louis-Mourier, Colombes
  - CHU Nantes, Nantes
  - Hospital Bichat-Hopitaux Universitaires Paris Nord Val de Seine, Paris
- Charite - Universitaetsmedizin Berlin, Berlin, Germany
- Italy (7):
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia BS
  - Azienda Sanitaria Ospedaliera Santa Croce E Carle - Cuneo, Cuneo CN
  - Ospedalle Galliera, Genova GE
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - U.O.C. Medicina Interna Azienda ospedaliero Universitaria Policlinico di Modena, Modena
  - IFO-San Gallicano IRCCS, Rome
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Materno-Infantile - Burlo Garofolo - Clinica Pediatrica, Trieste TS
- Japan (7):
  - Kobe University Hospital, Kobe, Hyōgo
  - Sophia Dermatology Clinic, Kanazawa, Ishikawa-ken
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Toyama University Hospital, Sugitani, Toyama
  - Mazda Hospital of Mazda Motor Corporation, Hiroshima
  - Hamamatsu University Hospital, Shizuoka
- Erasmus MC, Universitair Medisch Centrum Rotterdam, Rotterdam, Netherlands
- Haukeland University Hospital, Bergen, Norway
- Instytut hematologii i Transfuzjologii, Warsaw, Poland
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario, Madrid
  - Hospital General Universitario De Valencia, Valencia
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (4):
  - Salford Royal NHS Foundation Trust, Manchester, MN
  - St. John's Institute of Dermatology-Guy's & St Thomas' NHS Foundation Trust, London
  - Evelina London Children's Hospital - Guy's & St Thomas' NHS Foundation Trust, London
  - Southampton General Hospital - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No